CLINICAL TRIAL: NCT01446692
Title: Therapeutic Strategies for the Management of Patients With Major Depressive Disorder (MDD) and Suboptimal Response to Antidepressant Drugs in Primary Care: the Badalona Database Study
Brief Title: Badalona Major Depressive Disorder Database Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NES-XXX-2011/2
Record Dates: First submitted 2011-09-28; First posted 2011-10-05 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; primary care; real-world evidence; database
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with suboptimal response
- Patients with symptomatic remission

SUMMARY:
A retrospective study using a data base of anonymized medical records. The purpose of the study is to examine the different therapeutic strategies for the management of patients with major depressive disorder (MDD) and suboptimal response to antidepressant drugs in primary care

DETAILED DESCRIPTION:
Therapeutic strategies for the management of patients with major depressive disorder (MDD) and suboptimal response to antidepressant drugs in primary care: the Badalona database study

ELIGIBILITY:
Inclusion Criteria:

* An International Classification of Primary Care (ICPC-2) or DSM-IV-TR diagnosis for major depressive disorder (MDD)
* At least 8 weeks of antidepressant treatment during the identification period of 01 January 2008 - 31 December 2009
* 18 months of enrollment with medical and pharmacy records after index episode date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2260 (Actual)
Dates: Start 2011-11; Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Description of the antidepressant strategies switches | 18 months
  Number and type of treatment changes including combination, switch, or augmentation strategies.

SECONDARY OUTCOMES:
Health care resource utilization | 18 months
Health care costs | 18 months
Hamilton Depression Rating Scale | 18 months
Medication possession rate to evaluate adherence | 18 months
Referral to psychiatrist office | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Badalona, Spain